CLINICAL TRIAL: NCT02162615
Title: Restorelle® Transvaginal Mesh Versus Native Tissue Repair for Treatment of Pelvic Organ Prolapse, Restorelle 522 Study
Brief Title: Restorelle® Mesh Versus Native Tissue Repair for Prolapse
Status: Completed | Type: Observational
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: SU014
Record Dates: First submitted 2014-06-11; First posted 2014-06-13 (Estimated); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic Floor Disorder; Pelvic Organ Prolapse; Sexual Dysfunction; Mesh; POP; Transvaginal; Anterior; Posterior; Apical; Uterine Prolapse; Cystocele; Rectocele; Enterocele; Vaginal Vault Prolapse; Native Tissue Repair; Repair Augmented with Mesh; Pathological Conditions, Anatomical; Restorelle Direct Fix; Vaginal Mesh; Transvaginal Mesh
MeSH Terms: conditions — Pelvic Organ Prolapse; Pelvic Floor Disorders; Sexual Dysfunction, Physiological; Uterine Prolapse; Cystocele; Rectocele; Hernia; Pathological Conditions, Anatomical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Restorelle Direct Fix A: Anterior/Apical prolapse repair with Restorelle Direct Fix A
  Interventions: Device: Restorelle Direct Fix A
- Native Tissue Repair Anterior: Anterior/Apical prolapse repair with native tissue only
  Interventions: Procedure: Native Tissue Repair Anterior
- Restorelle Direct Fix P: Posterior/Apical prolapse repair with Restorelle Direct Fix P
  Interventions: Device: Restorelle Direct Fix P
- Native Tissue Repair Posterior: Posterior/Apical prolapse repair with native tissue only
  Interventions: Procedure: Native Tissue Repair Posterior

INTERVENTIONS:
Device: Restorelle Direct Fix A
  Groups: Restorelle Direct Fix A
Device: Restorelle Direct Fix P
  Groups: Restorelle Direct Fix P
Procedure: Native Tissue Repair Anterior
  Groups: Native Tissue Repair Anterior
Procedure: Native Tissue Repair Posterior
  Groups: Native Tissue Repair Posterior

SUMMARY:
The purpose of this study is to collect information on the safety and effectiveness of Restorelle Direct Fix mesh and the surgical procedure to implant Restorelle. These results will be compared to the safety and effectiveness results in patients who have native tissue repair (without mesh) as their pelvic organ prolapse treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female at least 18 years of age
* Subject has pelvic organ prolapse with leading edge at or beyond the hymen. At or beyond the hymen is defined as POP-Q scores of Ba ≥0 and C≥ -1/2 tvl or Bp ≥0 and C≥ -1/2 tvl
* Subject reports a bothersome bulge they can see or feel per PFDI-20 question 3, response of 2 or higher (i.e. responses of "somewhat", "moderately" or "quite a bit")
* Subject is willing to provide written informed consent
* Subject is willing and able to comply with the follow-up regimen

Exclusion Criteria:

* Subject is pregnant or intends to become pregnant during the study
* Subject has an active or chronic systemic infection including any gynecologic infection, untreated urinary tract infection (UTI), or tissue necrosis
* Subject has a history of pelvic organ cancer (e.g. uterine, ovarian, bladder, or cervical)
* Subject has had prior or is currently undergoing radiation, laser therapy, or chemotherapy in the pelvic area
* Subject has taken systemic steroids (within the last month), or immunosuppressive or immunomodulatory treatment (within the last 3 months)
* Subject has a systemic connective tissue disease (e.g. scleroderma, systemic lupus erythematosus (SLE), Marfan syndrome, Ehlers Danlos, collagenosis, polymyositis or polymyalgia rheumatica)
* Subject has chronic systemic pain that includes the pelvic area or chronic focal pain that involves the pelvis
* Subject has uncontrolled diabetes mellitus (DM)
* Subject has a known neurologic or medical condition affecting bladder function (e.g. multiple sclerosis, spinal cord injury, or stroke with residual neurologic deficit)
* Subject is seeking obliterative vaginal surgery as treatment for pelvic organ prolapse (colpocleisis)
* Subject is not able to conform to the modified dorsal lithotomy position
* Subject is currently participating in or plans to participate in another device or drug study during this study
* Subject has a known sensitivity to polypropylene
* Subject has had previous prolapse repair with mesh in the target compartment(s)
* Subject is planning to undergo a concomitant prolapse repair in a non-target compartment with anything other than native tissue repair

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female patients with pelvic organ prolapse who are candidates for transvaginal surgical repair.
Sampling Method: Non-Probability Sample
Enrollment: 810 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2021-11-06 (Actual)

PRIMARY OUTCOMES:
Recurrence of Prolapse | 12 Month
  Recurrent Prolapse measured anatomically at the target compartment by leading edge of prolapse beyond the hymenal ring by POP-Q examination, or additional surgical treatment for pelvic organ prolapse in the target vaginal compartment(s), or patient reporting symptoms of vaginal bulging.
Rate of device and procedure related serious adverse events | 12 Month

SECONDARY OUTCOMES:
Recurrence of Prolapse | 12 Month
  Recurrent prolapse is measured anatomically by leading edge of prolapse in the target compartment at or beyond the hymenal ring by POP-Q examination, or additional surgical treatment for pelvic organ prolapse in the target vaginal compartment(s), or patient reporting symptoms of vaginal bulging.
Recurrence of Prolapse | 36 Month
  Recurrent Prolapse is measured anatomically by leading edge of prolapse in the target compartment beyond the hymenal ring by POP-Q examination, or additional surgical treatment for pelvic organ prolapse in the target vaginal compartment(s), or patient reporting symptoms of vaginal bulging.
Recurrence of Prolapse | 36 Month
  Recurrent Prolapse measured anatomically by leading edge of prolapse in the target compartment at or beyond the hymenal ring by POP-Q examination, or additional surgical treatment for pelvic organ prolapse in the target vaginal compartment(s), or patient reporting symptoms of vaginal bulging.
Device or Procedure related AEs of interest | 36 months

OTHER OUTCOMES:
Additional adverse events | 36 months
Changes in Quality of Life scores for PFDI-20, PISQ-12, and PFIQ-7 | 36 months
Subjects experiencing vaginal bulge | 36 months
Rates of revision and/or re-surgery | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Paul Roovers, MD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (49):
- United States (33):
  - Sherry Thomas, M.D., Agoura Hills, California
  - Stanford University, Stanford, California
  - SurgOne Pelvic Solutions Center, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Center for Urogynecology and Pelvic Surgery, Christiana Care Health System, Newark, Delaware
  - MedStar Washington Hospital Center, National Center for Advanced Pelvic Surgery, Washington D.C., District of Columbia
  - Rosemark Women Care Specialists, Idaho Falls, Idaho
  - Andrew Shapiro, Owings Mills, Maryland
  - Baystate Health System, Springfield, Massachusetts
  - Female Pelvic Medicine & Urogynecology Institute of MI, Grand Rapids, Michigan
  - Beyer Research, Kalamazoo, Michigan
  - Adult & Pediatric Urology, PC, Omaha, Nebraska
  - Cooper University Hospital, Camden, New Jersey
  - Atlantic Health System, Morristown, New Jersey
  - Premier Medical Group of Hudson Valley, PC, Poughkeepsie, New York
  - Montefiore Medical Research Center, The Bronx, New York
  - Novant Health Urogynecology, Charlotte, North Carolina
  - Women's Pelvic Health and Continence Center, Hamlet, North Carolina
  - Novant Health Clinical Research, Winston-Salem, North Carolina
  - Akron Urogynecology Associates, Akron, Ohio
  - Good Samaritan Hospital, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - The Institute for Female Pelvic Medicine and Reconstructive Surgery, Allentown, Pennsylvania
  - Center for Women's Health of Lansdale, Lansdale, Pennsylvania
  - The Female Pelvic Health Center, Newtown, Pennsylvania
  - Wellspan Urogynecology and Pelvic Reconstructive Surgery, York, Pennsylvania
  - Sanford Research, Sioux Falls, South Dakota
  - Swan Urogynecology, Nashville, Tennessee
  - Central Texas Urogynecology and Continence Center, Austin, Texas
  - Scott D. Lauer, DO, PA, Colleyville, Texas
  - Carilion Clinic New River Valley, Christiansburg, Virginia
  - The Group for Women, Norfolk, Virginia
  - Integrity Medical Research, Mountlake Terrace, Washington
- Australia (2):
  - Centre for Advanced Reproductive Endosurgery, St Leonards, New South Wales
  - Mater Pelvic Health, Pimlico, Queensland
- UZ Leuven, Leuven, Belgium
- Canada (3):
  - Kingston General Hospital, Kingston, Ontario
  - Hôpital Maisonneuve-Rosemount, Montreal, Quebec
  - CHUS-CRC, Sherbrooke, Quebec
- France (2):
  - CHRU Lille, Lille
  - CHU Nimes, Nîmes
- Netherlands (8):
  - Bergman Clinics, Amsterdam
  - AMC Medical Center, Amsterdam
  - Bergman Clinics, Bilthoven
  - Amphia Hospital, Breda
  - Spaarne Gasthuis, Haarlem
  - Maastricht UMC, Maastricht
  - St. Antonius Ziekenhuis, Nieuwegein
  - ISALA, Zwolle

REFERENCES:
- [Derived] Sokol ER, Cosson M, Harris-Hicks JE, Mangel J, Thomas SL, Roovers JW. A Multicenter Prospective Study of Posterior Transvaginal Mesh Compared to Native Tissue Repair for Pelvic Organ Prolapse: 36 Month Outcomes. J Minim Invasive Gynecol. 2025 Oct;32(10):921-928. doi: 10.1016/j.jmig.2025.06.016. Epub 2025 Jun 26. PMID 40581283